CLINICAL TRIAL: NCT01988337
Title: Double Blind Randomized Controlled Clinical Trial of Lesion Progression After Treatment With Icon vs. Placebo in Caries Lesions in Young Adults Over 36 Months
Brief Title: Lesion Progression After Icon Treatment in Young Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slower than expected tooth decay in placebo group and insufficient recruitment.
Sponsor: DMG Dental Material Gesellschaft mbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TOPIC36
Record Dates: First submitted 2013-11-07; First posted 2013-11-20 (Estimated); Results first posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Caries; Salivary Function; Tooth Sensitivity
Keywords: Icon
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: Split-mouth design
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resin infiltration (Experimental): One proximal caries lesion (split mouth design) per patient will be treated using the resin infiltrant "Icon" (DMG, Hamburg, Germany) according to manufactures´ instructions.
  Interventions: Device: Resin infiltration
- Mock treatment (Sham Comparator): A second proximal caries lesion of each patient (split mouth design) will receive a placebo treatment to mimic "resin infiltration".
  Interventions: Other: Mock treatment

INTERVENTIONS:
Device: Resin infiltration — The study is a split-mouth design. One tooth with a proximal caries lesion will randomly receive the infiltrating resin (Icon) while the other will receive a placebo, according to the manufactures´ instruction for Icon. In short, teeth will be isolated with a rubber dam and the tooth surface cleaned with non-fluoride prophylactic paste and pumice. The Icon material will be applied following the manufacturer's instructions and light cured, followed by polished using interproximal finishing/polishing strips (Sof Lex, 3M ESPE, St Paul, MN). Subjects will be given a letter to take to their local dentist asking them not to treat the selected lesions without informing the investigator first.
  Other Names: Icon (DMG, Germany), approximal resin infiltration kit
  Arms: Resin infiltration
Other: Mock treatment — For the mock treatment the procedure will be identical to the "Resin Infiltration" intervention, with the exception that a placebo will be used. Essentially, syringes identical to the Icon materials will be supplied by DMG for the placebo procedure. The syringes will be filled with solutions having the same consistency and color as the Icon material.
  Arms: Mock treatment

SUMMARY:
This is a three year single site clinical evaluation of a FDA approved (510(k):K100062) lesion penetrating resin used to infiltrate and hamper progression of proximal carious lesions. The purpose of this study is to compare lesion progression infiltrated with (Icon, Hamburg, Germany) to a similar sized lesion in the same patient treated with a placebo. The study is designed as a randomized, controlled, prospective clinical trial with a three year follow-up evaluation period.

The clinical site will enroll 150 subjects (in the age range of 19 years or older) with 2 study lesions. The patients will be evaluated at six time points over a period of 3 years. Lesion status and caries risk will be monitored at 6-month intervals, while radiographic evaluation will be conducted at 12-month intervals at 1-, 2- and 3-year recall visits.

DETAILED DESCRIPTION:
Introduction Dental caries is the most widespread of all diseases. It causes destruction of tooth structure by dissolving the enamel on the outside of the tooth first and then progressing into the inside of the tooth. While it is possible to use traditional dental fillings to replace diseased tooth structure, it is far better to slow down or reverse the disease process so that no fillings are needed. One of the most difficult places to use preventive or non-surgical treatment is the contact area between teeth. Recently there is evolving interest in using composites to infiltrate enamel and dentin areas that have just begun to be destroyed by caries. The infiltration technique arrests the lesion progression by sealing the porous surface and restores the damage avoiding ongoing acidic damage of tooth structure.

Objective Assess the clinical efficacy s of using Icon to infiltrate initial lesions below the tooth surfaces that exist on the contact surfaces between posterior teeth as a means of stabilizing diseased tooth structure and arresting further lesion development.

Materials and Methods One hundred fifty volunteers (19+ years) with two early lesions in posterior teeth will be enrolled into a clinical trial to evaluate the clinical efficacy of infiltrating the lesions as compared to current watch-and-wait approaches that are combined with good oral hygiene and fluoride application. Each subject will have a treated lesion and a control lesion. Only small early lesions without clinical signs of surface cavitation will be selected. The control lesions will be stabilized through a normal preventive regimen, while the treatment lesions will be infiltrated with a resin. Lesion status will be monitored every six months by clinical examination and as well using annual radiographs.

Clinical Significance Infiltrating a caries lesion is a potential effective strategy to strengthen damaged tooth structure and to reduce caries progression without any surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Be age 19 years and older
* Have at least two vital carious teeth with caries ranging from enamel to just into dentin.

  * If the lesion is not on a 3rd molar
  * If the lesion is not developmental.
  * If the lesion is not cavitated
* Be a regular dental attendee able to return for assessments
* Be in good medical health and able to tolerate the dental procedure
* Have no chronic periodontitis which could compromise tooth retention.
* Have normal salivary function.
* Have normal bone levels
* No lingering cold sensitivity
* No periapical sensitivity
* No sensitivity to percussion

Exclusion Criteria:

* Do not meet the inclusion criteria
* Are not able to tolerate the time required for the study
* There is a history of an adverse reaction to any materials used in the study
* They are irregular dental attendees
* They maintain an unacceptable standard of oral hygiene.
* They have chronic periodontitis
* There is severe salivary gland dysfunction or reduced salivary flow is observed
* They are unable to return for recall appointments

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nate O. Lawson, Principal Investigator — Birmingham, Alabama 35294; US
Locations (1):
- University of Alabama, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from patients seeking treatment at the University of Alabama at Birmingham, School of Dentistry, USA, and through advertisements. The first participant was enrolled in August 2015 and the last was enrolled in August 2017.
Pre-assignment Details: Within-person study (split-mouth design): Per participant at least one lesion pair (two lesions on seperate teeth) were included. These two lesions were randomly allocated to either treatment (resin infiltration) or control (mock treatment) group resulting in paired lesions within the participants. For some participants more than one lesion pair was included.
Units Other Than Participants: Lesions
Groups:
- Resin Infiltration / Mock Treatment (Split-mouth; Participants With Paired Lesions): Within-person study (split-mouth design): For each participant at least one pair of lesions has been included, with one lesion per pair having been randomized to the treatment group (resin infiltration) and the other to the control group (mock treatment).
  Resin infiltration or Mock treatment was performed at baseline (study start) according to manufacturers' instructions for the respective study lesion; in addition to general caries preventive measures (standard-oral care hygiene treatment, diet counselling and fluoride regimen).
Period: Overall Study
Arm/Group | Resin Infiltration / Mock Treatment (Split-mouth; Participants With Paired Lesions)
Started | 56; 130 Lesions
Intervention (at Baseline) | 56; 130 Lesions (Received Resin Infiltration Treatment: 56 participants, 65 lesions Received Resin Mock (Control) Treatment: 56 participants, 65 lesions)
6 Months Follow up | 43; 102 Lesions (Followed up of those that received Resin Infiltration Treatment: 43 participants, 51 lesions Followed up of those that received Resin Mock (Control) Treatment: 43 participants, 51 lesions)
12 Months Follow up | 43; 102 Lesions (Followed up of those that received Resin Infiltration Treatment: 43 participants, 51 lesions Followed up of those that received Resin Mock (Control) Treatment: 43 participants, 51 lesions)
Completed (36 month follow up was expected for completion.) | 0; 0 Lesions
Not Completed | 56; 130 Lesions
Not completed — Study was terminated due to insufficient recruitment before 36 month follow up could be completed | 56

BASELINE CHARACTERISTICS:
Units Other Than Participants: Lesions
Groups:
- Resin Infiltration / Mock Treatment (Split-mouth; Participants With Paired Lesions): Within-person study (split-mouth design): For each participant at least one pair of lesions has been included, whereas one lesion per pair was randomized to the treatment group (resin infiltration) and the other to the control group (mock treatment).
  Resin infiltration or Mock treatment was performed at baseline (study start) according to manufacturers' instructions for the respective study lesion; in addition to general caries preventive measures (standard-oral care hygiene treatment, diet counselling and fluoride regimen).
Arm/Group | Resin Infiltration / Mock Treatment (Split-mouth; Participants With Paired Lesions)
Number analyzed (Participants) | 56
Number analyzed (Lesions) | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13
  Between 18 and 65 years | 43
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 30 [14 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 32
  Asian | 1
  African American | 19
  Hispanic or Latino | 3
  Two ethnicities (Asian and Hispanic) | 1
Region of Enrollment [Number; unit: participants]
  United States | 56
Caries Risk (CR) [Count of Participants; unit: Participants] — Caries risk (CR) was determined based on Bratthall/Petersson: Cariogram-a multifactorial risk assessment model for a multifactorial disease. Community Dent Oral Epidemiol. 2005 Aug: 33 (4): 256-64. The scale reaches from 0% (no risk) to 100% (high risk).
  Participants
    Low Caries Risk (CR<33%) | 17
    Moderate Caries Risk (34%<CR<66%) | 39
    High Caries Risk (67%<CR) | 0
Lesion size [Count of Units; unit: Lesions] — Categorical lesion depth as measured by radiographs. E1 (lesion within the outer half of enamel), E2 (inner half of enamel), D1 (outer third of dentin), D2 (middle third of dentin). Reference: Anusavice K. Present and future approaches for the control of caries. J Dent Educ. 2005;69(5):538-854. Population: In this within-person study (split-mouth design), at least one pair of lesions has been included per participant, with one lesion per pair being allocated to the treatment group (resin infiltration) and the other to the control group (mock treatment). Consequently, half of all study lesions belong to the treatment group and half to control group.
  Lesions
    number analyzed (Lesions) | 65
    Resin infiltration group: E1 | 40
    Resin infiltration group: E2 | 13
    Resin infiltration group: D1 | 12
    Resin infiltration group: D2 | 0
    Mock treatment group: E1 | 42
    Mock treatment group: E2 | 13
    Mock treatment group: D1 | 10
    Mock treatment group: D2 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Invasive Interventions (Fillings)
Description: Cumulative number of study lesions that have progressed to a state were an invasive intervention (filling) has been required to restore the teeth as determined via an dental examination (baseline versus 3 year follow up).
Time Frame: 3 years
Population: This study was terminated. The 3 year follow up was not reached for any enrolled participant at the time of termination.
Units Other Than Participants: Lesions
Groups:
- Resin Infiltration: Resin infiltration of lesion according to manufacturers instruction in addition to preventive measures (standard-oral care hygiene treatment, diet counselling and fluoride regimen).
- Mock Treatment: Mock treatment of lesion in addition to preventive measures (standard-oral care hygiene treatment, diet counselling and fluoride regimen).
Arm/Group | Resin Infiltration | Mock Treatment
Number analyzed (Participants) | 0 | 0
Number analyzed (Lesions) | 0 | 0

2. Secondary Outcome: Number of Lesions That Changed in Size (E1->E2->D1->D2-> Filling)
Description: Change in categorical lesion depth (progression to next depth category lesion; E1->E2->D1->D2->filling) as measured by pairwise comparison of radiographs (baseline versus follow up time point). E1 (lesion within the outer half of enamel), E2 (inner half of enamel), D1 (outer third of dentin), D2 (middle third of dentin). Reference: Anusavice K. Present and future approaches for the control of caries. J Dent Educ. 2005;69(5):538-854.
Time Frame: 6 months and 12 months
Population: The intended follow up time frame was 6, 12, 24 and 36 months. However, due to the termination of the study, only the 6 and 12 month follow ups were completed for the enrolled participants.
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Resin Infiltration | Mock Treatment
Number analyzed (Participants) | 43 | 43
Number analyzed (Lesions) | 51 | 51
Lesions
  Progressed lesions at 6 month follow up | 3 | 6
  Progressed lesions at 12 month follow up | 7 | 9

3. Other Pre Specified Outcome: Number of Lesions With Sensitivity to Percussion, Papillary Bleeding, Cold Response
Description: Teeth included in the study were clincially assed for sensitivity to percussion, papillary bleeding, cold response.
Time Frame: 6 months and 12 months
Population: as for outcome 2
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Resin Infiltration | Mock Treatment
Number analyzed (Participants) | 43 | 43
Number analyzed (Lesions) | 51 | 51
Lesions
  Papillary bleeding at 6 months | 19 | 18
  Papillary bleeding at 12 months | 4 | 4
  Cold response at 6 months | 1 | 0
  Cold response at 12 months | 0 | 1
  Sensitivity to percussion at 6 months | 0 | 0
  Sensitivity to percussion at 12 months | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline through 12 months.
Groups:
- Mock Treatment: Mock treatment of lesion according to manufacturers instruction in addition to preventive measures (standard-oral care hygiene treatment, diet counselling and fluoride regimen).
Arm/Group | Resin Infiltration | Mock Treatment
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 0/56 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT01988337/Prot_SAP_000.pdf